CLINICAL TRIAL: NCT00243295
Title: A Pilot Study to Validate the Feasibility of Injecting and Monitoring Recombinant Human Bone Morphogenetic Protein-2/Calcium Phosphate Matrix (rhBMP-2/CPM) in Subjects With Open Wedge Osteotomies
Brief Title: Study Evaluating rhMBP-2/CPM in Open Wedge Osteotomies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 3100N7-110
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2006-10

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; deformity of knee
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Drug: rhBMP-2/CPM

SUMMARY:
To assess the feasibility of using rhBMP-2/CPM in OWO as a surgical model for pharmacodynamic studies, with assessment of the following parameters:

* Injecting the desired volume of rhBMP-2/CPM within the defect
* Conducting longitudinal radiographic absorptiometry of the tibial defect in the presence of rhBMP-2/CPM.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 45 to 70 years of age
* Within 96 hours prior to dosing, the subject underwent a successful open wedge tibial osteotomy to correct medial compartment OA of the knee.
* Female subjects of childbearing potential must have a negative pregnancy test (hospital acceptable test), upon hospitalization for OWO and agree to use medically approved contraception for the duration of the study.

Other inclusion applies.

Exclusion Criteria:

* Subjects with pre-existing conditions of the knee or tibia that would confound an interpretation of results.
* Subjects for whom surgery in the opposite knee is planned during the 6 months of follow-up.
* Subjects with a history of malignancy or radiotherapy or chemotherapy for malignancy within the past 5 years, except subjects with a history of basal skin carcinoma.

Other exclusion applies.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Start 2003-11; Study Completion 2005-03

PRIMARY OUTCOMES:
Feasibility of injecting rhBMP-2/CPM using high tibial osteotomy as a surgical model for pharmacodynamic studies
Feasibility measures include
Injection of desired volume of rhBMP-2/CPM within the osteotomy defect
Ability to perform longitudinal radiographic absorptiometry of the defect in the presence of rhBMP-2/CPM.

SECONDARY OUTCOMES:
Safety of administering different volumes of rhBMP-2/CPM in high tibial osteotomy defects. Safety assessed by evaluation of adverse events reported during the duration of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer